CLINICAL TRIAL: NCT01663350
Title: Performance of the Verinata Health Prenatal Aneuploidy Test Compared to Current Fetal Aneuploidy Screening Results and Pregnancy Outcomes in an 'All-Risk' Population
Brief Title: Comparison of Aneuploidy Risk Evaluations
Acronym: CARE
Status: Completed | Type: Observational
Sponsor: Verinata Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VER-0007
Record Dates: First submitted 2012-07-31; First posted 2012-08-13 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Pregnancy; Down Syndrome; Edwards Syndrome; Patau Syndrome; Turners Syndrome
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All-risk pregnant women: All-risk pregnancies undergoing conventional forms of prenatal screening

SUMMARY:
This is a prospective, multi-center observational study designed to compare the test results of the Verinata Health Prenatal Aneuploidy Test to results of conventional prenatal screening for fetal chromosome abnormalities in 'all-risk' pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at enrollment
* Clinically confirmed pregnancy
* Gestational age ≥8 weeks, 0 days
* Planned or completed prenatal serum screening* (drawn during 1st and/or 2nd trimester)
* Pregnancy records accessible and available for data collection (e.g., results from screening, ultrasound examinations, invasive prenatal procedures if performed, and newborn hospital discharge exam)
* Able to provide consent for participation using language appropriate forms

Exclusion Criteria:

* Invasive prenatal procedure (amniocentesis or CVS) performed within 2 weeks prior to enrollment
* Prenatal screening determination by Nuchal Translucency (NT) measurement only

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of pregnant women at least 18 years of age, who meet the study eligibility criteria. Women who plan or have already completed prenatal screening for fetal aneuploidy during first and/or second trimester, will be recruited from approved participating clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Comparison of screen positive rates between investigational testing results and conventional screening results (standard of care). | 12 months
  The primary outcome of this study is the false positive rate of fetal aneuploidy detection for chromosome 21, 18, and 13 by the Verinata Health Prenatal Aneuploidy Test and screen positive rate for fetal trisomy (T21) and trisomy (T18) by conventional prenatal screening methods. Birth outcomes, or karyotype if available, will be used as the reference standard.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Sehnert, MD, Study Director — Verinata Health, Inc.
Locations (26):
- United States (26):
  - West Coast OB/GYN, San Diego, California
  - AD Williams Laboratory, Atlanta, Georgia
  - Prentice Women's Hospital, Chicago, Illinois
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Desert Perinatal Associates, Las Vegas, Nevada
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Virtua Perinatology Associates of Voorhees, Voorhees Township, New Jersey
  - Northshore University Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Lyndhurst Clinical Research, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Maternal Fetal Medicine, Cleveland, Ohio
  - MacDonald Clinical Research Unit, Mayfield Heights, Ohio
  - Network Office of Research and Innovation Lehigh Valley Health Network, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Clinical Research, Columbia, South Carolina
  - Greenville Hospital Systems, Greenville, South Carolina
  - Jackson Clinic, Jackson, Tennessee
  - Practice Research Organization, Dallas, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - The Group for Women, Norfolk, Virginia

REFERENCES:
- [Derived] Bianchi DW, Parker RL, Wentworth J, Madankumar R, Saffer C, Das AF, Craig JA, Chudova DI, Devers PL, Jones KW, Oliver K, Rava RP, Sehnert AJ; CARE Study Group. DNA sequencing versus standard prenatal aneuploidy screening. N Engl J Med. 2014 Feb 27;370(9):799-808. doi: 10.1056/NEJMoa1311037. PMID 24571752